CLINICAL TRIAL: NCT03322280
Title: TACE Combined With Iodine-125 Seeds Implantation Versus TACE Alone for Hepatocellular Carcinoma With Portal Vein Tumor Thrombus: A Prospective, Multicenter, Randomized, Controlled Study
Brief Title: TACE Combined With Iodine-125 Seeds Implantation for HCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: ZhuHai Hospital (Other); The First People's Hospital of Zhaoqing (Unknown); Foshan Sanshui District People's Hospital (Unknown); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Guangdong Provincial People's Hospital (Other); Sun Yat-sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIIR-01
Record Dates: First submitted 2017-06-09; First posted 2017-10-26 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Hepatocellular Carcinoma; Portal Vein Occlusion; Tumor Thrombus
Keywords: Hepatocellular carcinoma; Portal vein tumor thrombus; Transcatheter arterial chemoembolization; iodine-125 seed
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TACE+I-125 seeds (Experimental): TACE combined with iodine-125 seeds implantation
  Interventions: Procedure: TACE combined with iodine-125 seeds implantation
- TACE alone (Active Comparator): TACE alone
  Interventions: Procedure: TACE

INTERVENTIONS:
Procedure: TACE combined with iodine-125 seeds implantation — Conventional TACE with lipiodol was performed. Then Iodine-125 seed implantation into PVTT is conducted 7-10 days after TACE when liver function tests demonstrated values comparable to those obtained before TACE.
  Arms: TACE+I-125 seeds
Procedure: TACE — Only conventional TACE with lipiodol and chemotherapy drugs was performed.
  Arms: TACE alone

SUMMARY:
Portal vein tumour thrombus (PVTT) is a common complication of hepatocellular carcinoma (HCC). PVTT has a profound adverse effect on prognosis, with a very short median survival time (2-4 months). The presence of PVTT also limits treatment options, such as liver transplantation and curative resection. Although the Barcelona Clinic Liver Cancer group recommended sorafenib as a standard therapy for advanced-stage HCC, the optimal treatment for HCC with PVTT remains largely controversial.

Some studies have reported a survival benefit in patients with PVTT who underwent transarterial chemoembolization (TACE), even in patients with main portal vein (MPV) tumor thrombus. Iodine-125 brachytherapy had also showed promising efficacy as a new method for unresectable HCC with PVTT. Results of our previous study indicated that TACE combined with Iodine-125 seeds implantation might be a good choice for selected patients with PVTT. Thus, we conduct this study to farther evaluate the effect of TACE combined with Iodine-125 seeds implantation for HCC with PVTT.

270 patients with HCC and PVTT will be included and randomized to two group: group 1, patients received TACE combined with Iodine-125 seeds implantation; group 2, patients received TACE alone. TACE and Iodine-125 seeds implantation will be performed with a standardized procedure. Iodine-125 seeds implantation into PVTT (guided by CT) will be conducted 7 days after TACE.

All patients revisit our institutions for follow-up examinations including contrast enhanced CT/MRI and laboratory tests every 4-6 weeks after the first treatment. Patients who have a tumor response rating of complete response will be required to revisit 3 months interval. At each visit, TACE or Iodine-125 seeds implantation is repeated if the following criteria are reached: 1) images indicating viable intrahepatic tumor tissue or PVTT; 2) Child-Pugh class A or B, and no contraindication to TACE and Iodine-125 seeds implantation.

The primary end point of this study is overall survival. The secondary end points are time to tumor progression, disease control rate, duration of portal patency and adverse events. All adverse events are graded in accordance with Common Toxicity Criteria Adverse Events Version (CTCAE) 4.03.

DETAILED DESCRIPTION:
Background and purpose:

Hepatocellular carcinoma (HCC) is the 5th most common cancer in the world and the 3rd most prevalent cause of tumor-related deaths. Portal vein tumor thrombus (PVTT) occurs in up to 44% of HCC patients at the time of death and approximately 10-40% of patients at time of diagnosis. PVTT has a profound adverse effect on prognosis, with a very short median survival time (2-4 months). The presence of PVTT also limits treatment options, such as liver transplantation and curative resection. The optimal treatment for patients with HCC and PVTT remains largely controversial.

The Barcelona Clinic Liver Cancer (BCLC) group recommended the tyrosine kinase inhibitor sorafenib as a standard therapy for patients with advanced-stage HCC (BCLC stage C), including HCC patients with PVTT. However, in the Sorafenib Hepatocellular Carcinoma Assessment Randomized Protocol (SHARP) trail, on which the BCLC recommendations were based, patients with vascular invasion represented only 38.4% of the total study population. This result may not directly imply a survival gain with sorafenib treatment in HCC patients with PVTT. Additionally, the median survival time for patients with advanced HCC, including vascular invasion or extrahepatic metastases, treated with sorafenib is short - only 6.5 months in Asia. Thus, more effective treatment strategies have been strongly required to increase survival rate.

Some studies have reported a survival benefit in patients with PVTT who underwent transarterial chemoembolization (TACE), even in patients with main portal vein tumor thrombus. Iodine-125 brachytherapy alone had also showed promising efficacy as a new method for unresectable HCC with PVTT. Results of our previous study indicated that TACE combined with Iodine-125 seeds implantation might be a good choice for selected patients with PVTT. Thus, we conduct this study to farther evaluate the effect of TACE combined with Iodine-125 seeds implantation for HCC with PVTT.

Methods:

HCC was diagnosed by biopsy or according to the non-invasive criteria following the European Association for the Study of Liver/American Association for the study of Liver Disease guidelines. The presence of PVTT was confirmed by three-phase dynamic CT or MR. The types of PVTT were classified into four subgroups: type I, PVTT in segmental branches of portal vein or above; type II, PVTT affecting left/right portal vein; type III, PVTT affecting main portal vein (MPV); and type IV, PVTT affecting superior mesenteric vein (SMV).

270 patients met the eligibility criteria will be included in this study and randomized to two group: group 1, patients received TACE combined with Iodine-125 seeds implantation; group 2, patients received TACE alone.

TACE procedure:

solution of doxorubicin hydrochloride (20-40 mg) and 5-Fu (500-1000 mg) is infused into the feeder vessels of HCC. Then, An emulsion of 2-20 ml lipiodol and 20-50 mg lobaplatin is administered into the feeder vessels. The total amount of chemotherapy drugs is depended on the patient's body weight. Finally, gelatin sponge or polyvinyl alcohol (PVA) particles, which are mixed with contrast material, were administered into the feeder vessels until stasis of arterial flow was achieved. In patients with an arterioportal shunt, embolization with 300-1000 μm PVA is performed to occlude the shunt by superselective catheterization before infusion of lipiodol and lobaplatin emulsion.

Iodine-125 seeds implantation procedure:

Iodine-125 seeds implantation into PVTT is conducted 7 days after TACE when liver function tests demonstrated values comparable to those obtained before TACE. Each particle was 4.5 mm in length and 0.8 mm in diameter, with a radioactivity of 0.6-0.8mCi, radioactive half-life of 60.1days, and radiation energy of 27.4KeV. The volume and shape of PVTT is obtained by CT/MR images and used to calculate the matched peripheral dose and determine best percutaneous access route and numbers of Iodine-125 seeds using our three dimensional conformal radiation therapy Treatment Planning System (TPS). Implantation was guided by CT and Iodine-125 seeds are implanted into inside PVTT or around the PVTT (parenchymal or tumor issue from PVTT less than 1.7 cm) 5 mm apart along the length of PVTT using 18G needles.

Follow-up and re-treatment:

All patients revisit our institution for follow-up examinations including contrast enhanced CT/MRI every 4-6 weeks after the first treatment. The laboratory tests are checked within one week before and after the first TACE or Iodine-125 seed implantation, and every 4-6 weeks during follow-up. Patients who have a tumor response rating of complete response will be required to revisit 3 months interval. At each visit, TACE or Iodine-125 seed implantation or combination of TACE and Iodine-125 seed is repeated if the following criteria are reached: 1) images indicating viable intrahepatic tumor tissue or PVTT; 2) Child-Pugh class A or B, and no contraindication to TACE and Iodine-125 seeds implantation.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of HCC;
2. age between18 and 75 years;
3. type I PVTT, type II PVTT, or type III PVTT within 1.5cm extending in the main portal vein (if obstructive PVTT involve both the left and right portal vein or main portal vein, multiple collateral vessels are required);
4. Child-Pugh class A or B;
5. Eastern Cooperative Group performance status (ECOG) score of 0-2;
6. neutrophilic granulocyte count ≥ 1.5×10^9/L, platelet count ≥ 30×10^9/L, and hemoglobin level ≥ 85g/L;
7. serum bilirubin ≤ 51.3 μmol/L, albumin ≥ 28g/L, ALT and AST ≤ 5 times of the upper normal limit, and creatinine ≤ 20g/L;
8. prothrombin time ≤18s or international normalized ratio < 1.7.

Exclusion Criteria:

1. diffuse HCC;
2. extrahepatic metastasis;
3. obstructive PVTT involving both the left and right portal vein or main portal vein without collateral vessels,
4. type III PVTT affecting the main portal vein more than 1.5cm, or type IV PVTT;
5. previously surgery (resection or liver transplantation), local-regional therapies (e.g., radiofrequency ablation), intra-arterial chemoinfusion, TACE, radiotherapy, systemic chemotherapy, or molecular targeted drug therapy for HCC;
6. serious medical comorbidities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-09-18 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 24 months
  The time from date of randomization to death due to any cause.

SECONDARY OUTCOMES:
Adverse events | 24 months
  Side effects of TACE and iodine-125 seeds implantation were reported according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03
Progression free survival (PFS) | 24 months
  The time from randomization until the first occurrence of PD or death due to any cause, whichever occurs first.
Time to tumor progression (TTP) | 24 months
  The time from randomization until the date that disease progression (PD) was confirmed radiologically.
Objective response rate (ORR) | 24 months
  The percentage of patients who had a best overall tumor response rating of CR or PR.
Disease control rate (DCR) | 24 months
  Tumor response was evaluated with contrast-enhanced CT or MR imaging according to the modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria. Disease control rate was defined as the percentage of patients who had a best tumor response rating of complete response (CR), partial response (PR), or stable disease (SD), which was maintained for at least 4 weeks from the first manifestation of that modified Response Evaluation Criteria Solid Tumors rating.
Duration of portal patency | 24 months
  The time from randomization until the date that complete portal vein occlusion was confirmed (if the portal vein is patent at diagnosis).

CONTACTS AND LOCATIONS:
Overall Officials: Kangshun Zhu, MD, Study Chair — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The 2nd Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] El-Serag HB, Rudolph KL. Hepatocellular carcinoma: epidemiology and molecular carcinogenesis. Gastroenterology. 2007 Jun;132(7):2557-76. doi: 10.1053/j.gastro.2007.04.061. PMID 17570226
- [Background] Jemal A, Murray T, Ward E, Samuels A, Tiwari RC, Ghafoor A, Feuer EJ, Thun MJ. Cancer statistics, 2005. CA Cancer J Clin. 2005 Jan-Feb;55(1):10-30. doi: 10.3322/canjclin.55.1.10. PMID 15661684
- [Background] Pirisi M, Avellini C, Fabris C, Scott C, Bardus P, Soardo G, Beltrami CA, Bartoli E. Portal vein thrombosis in hepatocellular carcinoma: age and sex distribution in an autopsy study. J Cancer Res Clin Oncol. 1998;124(7):397-400. doi: 10.1007/s004320050189. PMID 9719503
- [Background] Cheung TK, Lai CL, Wong BC, Fung J, Yuen MF. Clinical features, biochemical parameters, and virological profiles of patients with hepatocellular carcinoma in Hong Kong. Aliment Pharmacol Ther. 2006 Aug 15;24(4):573-83. doi: 10.1111/j.1365-2036.2006.03029.x. PMID 16907890
- [Background] Minagawa M, Makuuchi M. Treatment of hepatocellular carcinoma accompanied by portal vein tumor thrombus. World J Gastroenterol. 2006 Dec 21;12(47):7561-7. doi: 10.3748/wjg.v12.i47.7561. PMID 17171782
- [Background] Llovet JM, Bustamante J, Castells A, Vilana R, Ayuso Mdel C, Sala M, Bru C, Rodes J, Bruix J. Natural history of untreated nonsurgical hepatocellular carcinoma: rationale for the design and evaluation of therapeutic trials. Hepatology. 1999 Jan;29(1):62-7. doi: 10.1002/hep.510290145. PMID 9862851
- [Background] Schoniger-Hekele M, Muller C, Kutilek M, Oesterreicher C, Ferenci P, Gangl A. Hepatocellular carcinoma in Central Europe: prognostic features and survival. Gut. 2001 Jan;48(1):103-9. doi: 10.1136/gut.48.1.103. PMID 11115830
- [Background] Omata M, Lesmana LA, Tateishi R, Chen PJ, Lin SM, Yoshida H, Kudo M, Lee JM, Choi BI, Poon RT, Shiina S, Cheng AL, Jia JD, Obi S, Han KH, Jafri W, Chow P, Lim SG, Chawla YK, Budihusodo U, Gani RA, Lesmana CR, Putranto TA, Liaw YF, Sarin SK. Asian Pacific Association for the Study of the Liver consensus recommendations on hepatocellular carcinoma. Hepatol Int. 2010 Mar 18;4(2):439-74. doi: 10.1007/s12072-010-9165-7. PMID 20827404
- [Background] Forner A, Reig ME, de Lope CR, Bruix J. Current strategy for staging and treatment: the BCLC update and future prospects. Semin Liver Dis. 2010 Feb;30(1):61-74. doi: 10.1055/s-0030-1247133. Epub 2010 Feb 19. PMID 20175034
- [Background] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Background] Llovet JM, Bru C, Bruix J. Prognosis of hepatocellular carcinoma: the BCLC staging classification. Semin Liver Dis. 1999;19(3):329-38. doi: 10.1055/s-2007-1007122. PMID 10518312
- [Background] Pinter M, Hucke F, Graziadei I, Vogel W, Maieron A, Konigsberg R, Stauber R, Grunberger B, Muller C, Kolblinger C, Peck-Radosavljevic M, Sieghart W. Advanced-stage hepatocellular carcinoma: transarterial chemoembolization versus sorafenib. Radiology. 2012 May;263(2):590-9. doi: 10.1148/radiol.12111550. Epub 2012 Mar 21. PMID 22438359
- [Background] Chung GE, Lee JH, Kim HY, Hwang SY, Kim JS, Chung JW, Yoon JH, Lee HS, Kim YJ. Transarterial chemoembolization can be safely performed in patients with hepatocellular carcinoma invading the main portal vein and may improve the overall survival. Radiology. 2011 Feb;258(2):627-34. doi: 10.1148/radiol.10101058. PMID 21273524
- [Background] Lee HS, Kim JS, Choi IJ, Chung JW, Park JH, Kim CY. The safety and efficacy of transcatheter arterial chemoembolization in the treatment of patients with hepatocellular carcinoma and main portal vein obstruction. A prospective controlled study. Cancer. 1997 Jun 1;79(11):2087-94. PMID 9179054
- [Background] Luo J, Guo RP, Lai EC, Zhang YJ, Lau WY, Chen MS, Shi M. Transarterial chemoembolization for unresectable hepatocellular carcinoma with portal vein tumor thrombosis: a prospective comparative study. Ann Surg Oncol. 2011 Feb;18(2):413-20. doi: 10.1245/s10434-010-1321-8. Epub 2010 Sep 14. PMID 20839057
- [Background] Xue TC, Xie XY, Zhang L, Yin X, Zhang BH, Ren ZG. Transarterial chemoembolization for hepatocellular carcinoma with portal vein tumor thrombus: a meta-analysis. BMC Gastroenterol. 2013 Apr 8;13:60. doi: 10.1186/1471-230X-13-60. PMID 23566041
- [Background] Zhang FJ, Li CX, Jiao DC, Zhang NH, Wu PH, Duan GF, Wu YX. CT guided 125iodine seed implantation for portal vein tumor thrombus in primary hepatocellular carcinoma. Chin Med J (Engl). 2008 Dec 5;121(23):2410-4. PMID 19102958
- [Background] Huang M, Lin Q, Wang H, Chen J, Bai M, Wang L, Zhu K, Jiang Z, Guan S, Li Z, Qian J, Li M, Pang P, Shan H. Survival benefit of chemoembolization plus Iodine125 seed implantation in unresectable hepatitis B-related hepatocellular carcinoma with PVTT: a retrospective matched cohort study. Eur Radiol. 2016 Oct;26(10):3428-36. doi: 10.1007/s00330-015-4198-x. Epub 2016 Jan 20. PMID 26792430
- [Background] Shi J, Lai EC, Li N, Guo WX, Xue J, Lau WY, Wu MC, Cheng SQ. A new classification for hepatocellular carcinoma with portal vein tumor thrombus. J Hepatobiliary Pancreat Sci. 2011 Jan;18(1):74-80. doi: 10.1007/s00534-010-0314-0. PMID 20686792